CLINICAL TRIAL: NCT05607992
Title: Brief Internet-delivered Exposure-based Therapy to Reduce Post-traumatic Stress Symptoms and Cardiac Anxiety After Acute Coronary Syndrome: a Pilot Randomized Clinical Trial
Brief Title: Brief Internet-delivered CBT After ACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Columbia University (Other)
Responsible Party: Principal Investigator, Josefin Särnholm, Principal Investigator, PhD, Lic. psychologist, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P30AG064198 (NIH)
Record Dates: First submitted 2022-10-27; First posted 2022-11-07 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Psychological Trauma; Acute Coronary Syndrome
Keywords: Acute coronary syndrome; Posttraumatic stress disorder; Cardiac anxiety; Cognitive behavioral therapy
MeSH Terms: conditions — Psychological Trauma; Acute Coronary Syndrome; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief exposure-based CBT (Experimental): * Patient education: Common reactions following ACS. The role of PTS, cardiac anxiety and avoidance behavior on quality of life and physical health and health behaviors.
  * Labeling i.e., describe cardiac-related symptoms, thoughts, and feelings.
  * Imaginal exposure to reduce PTSS: Imaginal processing and revisiting of the memory of the ACS
  * Interoceptive exposure to physical sensations (e.g., palpitations due to physical activity) to reduce fear of these symptoms.
  * Gradual exposure in-vivo to avoided situations, activities and physical activity. Continuously use labeling while conducting exposure exercises.
  * Relapse prevention: Prevention of relapse into avoidance behaviors by identifying risk situations and encouragement of maintaining a healthy physically active lifestyle.
  Interventions: Behavioral: Brief exposure-based CBT
- Waitlist control (No Intervention): The waitlist control will be offered an opportunity to participate in the intervention after the 2-month intervention evaluation period.

INTERVENTIONS:
Behavioral: Brief exposure-based CBT — The 5-week intervention is psychologist-guided and delivered via text-based interactive online treatment modules, where patients complete weekly homework assignments and have regular online contact with psychologists with training in CBT for cardiac disease. Key components include imaginal exposure of the ACS event, interoceptive exposure through at home physical activity that stimulats the CV system, exposure in-vivo to reduce avoided situations, and activities to enhance physical activity wellbeing. Labeling (i.e., describing cardiac-related symptoms, thoughts, and feelings) will be used continuously during treatment to enhance the effect of exposure.
  Arms: Brief exposure-based CBT

SUMMARY:
The purpose of the present pilot study is to evaluate the feasibility and potential efficacy of a brief, internet-delivered CBT protocol provided early after acute coronary syndrome (ACS).

DETAILED DESCRIPTION:
Acute coronary syndrome (ACS; myocardial infarction (MI) or unstable angina (UA)) is one of the leading causes of mortality and health loss globally. ACS is a stressful and potentially life-threatening cardiovascular event, and many patients develop symptoms of post-traumatic stress (PTSS) and cardiac anxiety post ACS, which have been shown to negatively affect patients' long-term cardiovascular prognosis.The aim of the proposed pilot study is to develop and evaluate a brief internet-delivered exposure-based CBT intervention provided early following ACS to reduce ACS-related PTSS, cardiac anxiety. and increase physical activity and quality of life. Patients with recent ACS (≥ 4 weeks to 6 months) and with elevated PTSS and anxiety will be eligible. After informed consent, patients will be randomized to internet-delivered CBT (N=15) or to a wait-list control group (N=15). The treatment is a 5 week, therapist-guided, internet-delivered intervention which includes imaginal exposure, interoceptive exposure, and exposure in-vivo. Assessments will be conducted at baseline, immediate post-treatment, and 2- and 6- months after treatment. The wait-list will be crossed over to CBT after completion of the 2 month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* (A) ACS ≥ four weeks to six months before assessment (MI type 1 STEMI/NSTEMI and UA)
* (B) Age 18-80 years
* (C) Symptoms of PTSD and/or cardiac anxiety that leads to distress and/or interferes with daily life (PCL5; ≥ 10, CAQ: ≥20)
* (D) On standard of care medical treatment for the cardiac condition according to Swedish cardiovascular guidelines
* (E) Ability to read and write in Swedish.

Exclusion Criteria:

* (F) Heart failure with severe systolic dysfunction (ejection fraction ≤ 35%)
* (G) Significant valvular disease
* (H) Planned coronary artery bypass surgery or percutaneous interventions
* (I) Any medical restriction to physical exercise
* (J) Severe uncontrolled medical illness i.e., advanced cancer
* (K) Grade 3 hypertension (i.e., blood pressure ≥ 180 systolic and/or 110 diastolic)
* (L) Severe psychiatric disorder, active suicidal ideations or cognitive impairment that precludes provision of informed consent or study activities
* (M) Alcohol dependency
* (N) Ongoing psychological treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-05-18 (Actual); Primary Completion 2024-08-21 (Actual); Study Completion 2024-08-21 (Actual)

PRIMARY OUTCOMES:
Seattle Angina Questionnaire | Baseline to 3 months
  A measure of coronary artery disease on five scales: physical limitation scale, anginal stability scale, anginal frequency scale, treatment satisfaction scale, and the disease perception scale. With a score ranging from 0 to 100. A higher score indicating a better quality of life.
Acceptability: Client satisfaction Questionnaire | Baseline to 5 weeks
  Treatment satisfaction, score ranging from 0 to 32, with a higher score indication more satisfaction with the treatment.
Percentage of enrolled participants who complete the treatment | Baseline to 5 weeks
  Feasibility of the intervention components will be assessed by >60% assessed as treatment completers. Descriptive analysis will also provide number of messages and therapist time.
Adverse events | Baseline to 5 weeks
  Potential adverse reactions to the treatment. Participants will be asked to report and rate the short- and long term discomfort of the adverse event on a scale from 0 ('did not affect me at all') and 3 ('affected me very negatively').

SECONDARY OUTCOMES:
Seattle Angina Questionnaire | Baseline to 5 weeks
  A measure of coronary artery disease on five scales: physical limitation scale, anginal stability scale, anginal frequency scale, treatment satisfaction scale, and the disease perception scale. With a score ranging from 0 to 100. A higher score indicating a better quality of life.
Seattle Angina Questionnaire | Baseline to 7 months
  A measure of coronary artery disease on five scales: physical limitation scale, anginal stability scale, anginal frequency scale, treatment satisfaction scale, and the disease perception scale. With a score ranging from 0 to 100. A higher score indicating a better quality of life.
Seattle Angina Questionnaire | Change over 5 measurement points measured from baseline and weekly for 5 weeks during treatment
  A measure of coronary artery disease on five scales: physical limitation scale, anginal stability scale, anginal frequency scale, treatment satisfaction scale, and the disease perception scale. With a score ranging from 0 to 100. A higher score indicating a better quality of life.
The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5 | Baseline to 5 weeks
  Measure of post traumatic stress, score ranging from 0-80, with a higher score indicating more post traumatic stress.
The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5 | Baseline to 3 months
  Measure of post traumatic stress, score ranging from 0-80, with a higher score indicating more post traumatic stress.
The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5 | Baseline to 7 months
  Measure of post traumatic stress, score ranging from 0-80, with a higher score indicating more post traumatic stress.
The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5 | Change over 5 measurement points measured from baseline and weekly for 5 weeks during treatment
  Measure of post traumatic stress, score ranging from 0-80, with a higher score indicating more post traumatic stress.
Cardiac anxiety questionnaire | Baseline to 5 weeks
  Measure of cardiac anxiety, fear, avoidance and attention. The score ranges between 0 and 72, with a greater score indicating elevated cardiac anxiety.
Cardiac anxiety questionnaire | Baseline to 3 months
  Measure of cardiac anxiety, fear, avoidance and attention. The score ranges between 0 and 72, with a greater score indicating elevated cardiac anxiety.
Cardiac anxiety questionnaire | Baseline to 7 months
  Measure of cardiac anxiety, fear, avoidance and attention. The score ranges between 0 and 72, with a greater score indicating elevated cardiac anxiety.
Cardiac anxiety questionnaire | Change over 5 measurement points measured from baseline and weekly for 5 weeks during treatment
  Measure of cardiac anxiety, fear, avoidance and attention. The score ranges between 0 and 72, with a greater score indicating elevated cardiac anxiety.
Myocardial infarction behavior questionnaire | Baseline to 8 weeks.
  MI-related avoidance questionnaire behaviors developed by the research group. score ranging from 0 to 68 . Higher scores indicate more avoidance behavior.
Myocardial infarction behavior questionnaire | Baseline to 3 months
  MI-related avoidance questionnaire behaviors developed by the research group. score ranging from 0 to 68 . Higher scores indicate more avoidance behavior.
Myocardial infarction behavior questionnaire | Baseline to 7 months
  MI-related avoidance questionnaire behaviors developed by the research group. score ranging from 0 to 68 . Higher scores indicate more avoidance behavior.
Body Sensation Questionnaire | Baseline to 8 weeks
  Fear of bodily symptoms, score ranging from 0 to 72 . Higher scores indicate more fear of body sensations.
Body Sensation Questionnaire | Baseline to 3 months
  Fear of bodily symptoms, score ranging from 0 to 72 . Higher scores indicate more fear of body sensations.
Body Sensation Questionnaire | Baseline to 7 months
  Fear of bodily symptoms, score ranging from 0 to 72 . Higher scores indicate more fear of body sensations.
Symptom checklist Severity and Frequency Scale (SCL, adapted to coronary artery disease) | Baseline to 8 weeks.
  Cardiac-related symptoms in two sub scales A) frequency: score ranging from 0-48, with higher score indicating higher frequency of symptoms, B) severity of experienced symptom: score ranging from 0- 48, with a higher score indicating more severe symptoms
Symptom checklist Severity and Frequency Scale (SCL, adapted to coronary artery disease) | Baseline to 3 months
  Cardiac-related symptoms in two sub scales A) frequency: score ranging from 0-48, with higher score indicating higher frequency of symptoms, B) severity of experienced symptom: score ranging from 0- 48, with a higher score indicating more severe symptoms
Symptom checklist Severity and Frequency Scale (SCL, adapted to coronary artery disease) | Baseline to 7 months
  Cardiac-related symptoms in two sub scales A) frequency: score ranging from 0-48, with higher score indicating higher frequency of symptoms, B) severity of experienced symptom: score ranging from 0- 48, with a higher score indicating more severe symptoms
12-Item Short-Form Health Survey | Baseline to 5 weeks
  General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life
12-Item Short-Form Health Survey | Baseline to 3 months
  General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life
12-Item Short-Form Health Survey | Baseline to 7 months
  General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life
Patient Health Questionnaire-9 | Baseline to 5 weeks
  Measure of depression, score ranging 0 to 27 with a higher score indicating higher level of depression
Patient Health Questionnaire-9 | Baseline to 3 months
  Measure of depression, score ranging 0 to 27 with a higher score indicating higher level of depression
Patient Health Questionnaire-9 | Baseline to 7 months
  Measure of depression, score ranging 0 to 27 with a higher score indicating higher level of depression
Generalized Anxiety Disorder 7-item | Baseline to 5 weeks.
  General anxiety, score ranging from 0-21, with a higher score indicating more anxiety and worry.
Generalized Anxiety Disorder 7-item | Baseline to 3 months
  General anxiety, score ranging from 0-21, with a higher score indicating more anxiety and worry.
Generalized Anxiety Disorder 7-item | Baseline to 7 months
  General anxiety, score ranging from 0-21, with a higher score indicating more anxiety and worry.
Perceived stress scale 4-item | Baseline to 5 weeks
  Stress reactivity. A greater score indicate more perceived stress.
Perceived stress scale 4-item | Baseline to 3 months
  Stress reactivity. A greater score indicate more perceived stress.
Perceived stress scale 4-item | Baseline to 7 months
  Stress reactivity. A greater score indicate more perceived stress.
The Godin Leisure-time Exercise and International Physical Activity Questionnaire 1 item on inactivity | Baseline to 5 weeks
  Level of physical activity and inactivity: On the Godin leisure-time excercise: The participant rate numbers of time per week that they engage in physical activity. The numb ers are the categorized in to low, moderate, and high levels of physical activity. And from International Physical Activity Questionnaire we will use 1 item on inactivity
The Godin Leisure-time Exercise and International Physical Activity Questionnaire 1 item on inactivity | Baseline to 3 months
  Level of physical activity and inactivity: On the Godin leisure-time excercise: The participant rate numbers of time per week that they engage in physical activity. The numb ers are the categorized in to low, moderate, and high levels of physical activity. And from International Physical Activity Questionnaire we will use 1 item on inactivity
The Godin Leisure-time Exercise and International Physical Activity Questionnaire 1 item on inactivity | Baseline to 7 months
  Level of physical activity and inactivity: On the Godin leisure-time excercise: The participant rate numbers of time per week that they engage in physical activity. The numb ers are the categorized in to low, moderate, and high levels of physical activity. And from International Physical Activity Questionnaire we will use 1 item on inactivity
Lifestyle factors: The national Board of health and Welfare questionnaire | Baseline to 8 weeks
  Questionnaire regarding diet (5 item), tobacco (2 item) and alcohol (3 item) diet (5 item), tobacco (2 item) and alcohol (3 item)
Lifestyle factors: The national Board of health and Welfare questionnaire | Baseline to 3 months
  Questionnaire regarding diet (5 item), tobacco (2 item) and alcohol (3 item) diet (5 item), tobacco (2 item) and alcohol (3 item)
Lifestyle factors: The national Board of health and Welfare questionnaire | Baseline to 7 months
  Questionnaire regarding diet (5 item), tobacco (2 item) and alcohol (3 item) diet (5 item), tobacco (2 item) and alcohol (3 item)
University of Toronto Atrial fibrillation Severity Scale (AFSS) | Baseline to 5 weeks
  3 item on cardiac-specific healthcare consumption. Scores ranges 0-15 with a higher score indicating more cardiac-related healthcare consumption.
University of Toronto Atrial fibrillation Severity Scale (AFSS) | Baseline to 3 months
  3 item on cardiac-specific healthcare consumption. Scores ranges 0-15 with a higher score indicating more cardiac-related healthcare consumption.
University of Toronto Atrial fibrillation Severity Scale (AFSS) | Baseline to 7 months
  3 item on cardiac-specific healthcare consumption. Scores ranges 0-15 with a higher score indicating more cardiac-related healthcare consumption.

OTHER OUTCOMES:
Adverse events | Baseline to 3 months
  Potential adverse reactions to the treatment. Participants will be asked to report and rate the short- and long term discomfort of the adverse event on a scale from 0 ('did not affect me at all') and 3 ('affected me very negatively').
Adverse events | Baseline to 7 months
  Potential adverse reactions to the treatment. Participants will be asked to report and rate the short- and long term discomfort of the adverse event on a scale from 0 ('did not affect me at all') and 3 ('affected me very negatively').
Adverse events | 5 measurement points measured from baseline and weekly for 5 weeks during treatment
  Potential adverse reactions to the treatment. Participants will be asked to report and rate the short- and long term discomfort of the adverse event on a scale from 0 ('did not affect me at all') and 3 ('affected me very negatively').
AFFS/SCL-4 | Change over 5 measurement points measured from baseline and weekly for 8 weeks during treatment ]
  4 items derived from the Symptoms Checklist (SCL) and the Atrial Fibrillation Severity Scale (AFSS) measuring disabling cardiac symptoms

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Karolinska University Hospital, Stockholm
  - Karolinska Institutet, Stockholm

IPD SHARING:
Plan to Share IPD: No